CLINICAL TRIAL: NCT05093309
Title: Preventing Opioid Overdose Deaths by Empowering Pharmacists to Dispense Naloxone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lindsey Hohmann, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R36HS026669-01A1 (AHRQ)
Record Dates: First submitted 2021-10-04; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Opioid Overdose
Keywords: naloxone; community pharmacy; implementation
MeSH Terms: conditions — Opiate Overdose | interventions — Health Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group received naloxone resources + monthly reminders + educational webinar.
  Interventions: Behavioral: Educational Webinar; Behavioral: Resources; Behavioral: Reminders
- Control (No Intervention): The control group received naloxone resources + monthly reminders + delayed educational webinar (after the 3-month study period).

INTERVENTIONS:
Behavioral: Educational Webinar — At month 1 of the study period, the educational webinar was presented by expert speakers and consisted of 3 modules: 1) naloxone basics; 2) naloxone service implementation strategies; and 3) naloxone recommendation communication strategies. Participants were mailed naloxone nasal spray and auto-injector training devices prior to attending the online webinar so that they could follow along during demonstrations.
  Other Names: Empowering Community Pharmacists Webinar
  Arms: Intervention
Behavioral: Resources — After completing the baseline survey, both control and intervention groups were provided with a basic publicly available flyer about naloxone dosage forms in order to ensure all participants could provide adequate patient care.
  Other Names: Flyers
  Arms: Intervention
Behavioral: Reminders — Reminders consisted of monthly emails from investigators for the purpose of retaining study engagement.
  Other Names: Nudge
  Arms: Intervention

SUMMARY:
Objectives: The purpose of this study was to assess the impact of the Empowering Community Pharmacists program on pharmacists' knowledge, perceived barriers, attitudes, confidence, and intentions regarding naloxone services implementation, as well as change in number of naloxone prescriptions dispensed.

Methods: A 3-month pragmatic randomized controlled trial was conducted in 2018-2019. Alabama community pharmacists were recruited by email, phone, fax, and mailed postcards and randomized to intervention (monthly resources/reminders + educational webinar) or control (monthly resources/reminders + delayed educational webinar). Outcome measures were assessed via online surveys at baseline (T1), immediately post-intervention (T2), and 3-months post-intervention (T3), including: naloxone knowledge (percent correct); perceived barriers, attitudes, and confidence regarding naloxone services implementation (7-point Likert-type scale, 1=strongly disagree to 7=strongly agree); and number of naloxone prescriptions dispensed. Mean differences between control and intervention groups from T1-T3 were assessed using two-way mixed ANOVA and adjusted analyses were conducted using generalized estimating equations (GEE) with negative binomial distribution (alpha=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Registered pharmacists.
* Employed at least 30 hours per week at a community pharmacy.
* Employed at a community pharmacy located in one of 20 Alabama priority counties with the highest opioid overdose mortality rates.

Exclusion Criteria:

* Multiple pharmacists from the same pharmacy site.
* Members of the stakeholder panel (from the formative phase of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Change in naloxone knowledge from baseline to immediately post-intervention and 3 months post-intervention | 3 months: baseline (T1), immediately post-intervention (T2), and 3 months post-intervention (T3)
  Knowledge about naloxone was measured via online survey. Knowledge was measured as percent correct on a 7-item index adapted from Williams' (2013) Opioid Overdose Knowledge Scale (OOKS).
Change in perceived barriers from baseline to immediately post-intervention and 3 months post-intervention | 3 months: baseline (T1), immediately post-intervention (T2), and 3 months post-intervention (T3)
  Perceived barriers to adoption/implementation of pharmacy-based naloxone services was measured via online survey. Barriers (20-items) were measured using 7-point Likert-type scales (1=strongly disagree, 7=strongly agree) and informed by Nielsen et al (2016) and Williams' (2013) Opioid Overdose Attitude Scale (OOAS).
Change in attitudes from baseline to immediately post-intervention and 3 months post-intervention | 3 months: baseline (T1), immediately post-intervention (T2), and 3 months post-intervention (T3)
  Attitudes regarding pharmacy-based naloxone services was measured via online survey. Attitudes (15-items) were measured using 7-point Likert-type scales (1=strongly disagree, 7=strongly agree) and informed by Nielsen et al (2016) and Williams' (2013) Opioid Overdose Attitude Scale (OOAS).
Change in confidence from baseline to immediately post-intervention and 3 months post-intervention | 3 months: baseline (T1), immediately post-intervention (T2), and 3 months post-intervention (T3)
  Confidence in performing naloxone dispensing behaviors was measured via online survey. Confidence (10-items) was measured using 7-point Likert-type scales (1=strongly disagree, 7=strongly agree) and informed by Nielsen et al (2016) and Williams' (2013) Opioid Overdose Attitude Scale (OOAS).
Change in intention from baseline to immediately post-intervention and 3 months post-intervention | 3 months: baseline (T1), immediately post-intervention (T2), and 3 months post-intervention (T3)
  Intention to dispense naloxone or perform naloxone services in the next three months was measured via online survey. The 5-item intention construct was measured using a 7-point Likert-type scale from 1=strongly disagree to 7=strongly agree and informed by an existing intention measure by Urmie et al (2007).

SECONDARY OUTCOMES:
Change in number of naloxone prescriptions dispensed from baseline to 3 months post-intervention | 3 months: baseline (T1) and 3 months post-intervention (T3)
  The number of naloxone prescriptions dispensed over 3 months before and after the intervention was assessed via self-report at T1 and T3. Participants utilized national drug codes (NDCs) within their pharmacy dispensing software to identify naloxone dispensing information.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Hohmann, PharmD, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University Harrison School of Pharmacy, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
In order to protect confidentiality of participants, data will not be shared.

REFERENCES:
- [Derived] Hohmann LA, Fox BI, Garza KB, Wang CH, Correia C, Curran GM, Westrick SC. Impact of a Multicomponent Educational Intervention on Community Pharmacy-Based Naloxone Services Implementation: A Pragmatic Randomized Controlled Trial. Ann Pharmacother. 2023 Jun;57(6):677-695. doi: 10.1177/10600280221120405. Epub 2022 Sep 1. PMID 36047381